CLINICAL TRIAL: NCT07230509
Title: Efficacy of Pancreatic Parenchymal N-Butyl-2-Cyanoacrylate Injection in Pancreaticojejunostomy After Pancreaticoduodenectomy: A Randomized Controlled Trial
Brief Title: Pancreatic Parenchymal Injection of N-butyl-2-cyanoacrylate
Acronym: NBCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1703/09/2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreaticoduodenectomy; Postoperative Pancreatic Fistula; Pancreas Cancer; Periampullary Cancer
Keywords: Pancreatic surgery; Anastomotic leak; Tissue adhesive; Postoperative Pancreatic Fistula (POPF); Pancreaticoduodenectomy (PD); Pancreaticojejunostomy (PJ)
MeSH Terms: conditions — Pancreatic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: Patients randomized to the groups will receive a standardized volume (e.g., 0.5 mL of a 1:1 mixture of NBCA and Lipiodol) of N-Butyl-2-Cyanoacrylate injected into the pancreatic parenchyma during pancreaticojejunostomy. The injection will be performed using a fine-gauge needle at multiple points to ensure even distribution. The specific NBCA product will be a commercially available, cyanoacrylate adhesive (e.g., Histoacryl®).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-butyl-2-cyanoacrylate (Histoacryl® )Injection Group. (Experimental): Patients randomized to this group will undergo pancreaticoduodenectomy and pancreaticojejunostomy with pancreatic parenchymal injection of N-butyl-2-cyanoacrylate during pancreaticoduodenectomy.
  Interventions: Drug: Pancreatic parenchymal injection of N-butyl-2- cyanoacrylate(Histoacryl®)Injection Group.
- Standard Pancreaticojejunostomy (Active Comparator): Patients randomized to this group will undergo pancreaticoduodenectomy and pancreaticojejunostomy using the standard surgical technique of the institution, without the application of N-Butyl-2-Cyanoacrylate or any other sealant to the pancreatic anastomosis. No placebo injection will be administered.
  Interventions: Procedure: Standard Pancreaticojejunostomy

INTERVENTIONS:
Drug: Pancreatic parenchymal injection of N-butyl-2- cyanoacrylate(Histoacryl®)Injection Group. — This procedure is integrated into the standard pancreaticoduodenectomy. Injection of Histoacryl® (n-butyl-2-cyanoacrylate) mixed with Lipiodol® (1:1 ratio) into the pancreatic parenchyma circumferentially (3, 6, 9, and 12 o'clock positions) around the main pancreatic duct (MPD) orifice, extending 5-8 mm deep and 5-10 mm laterally from the future anastomotic line, avoiding the main pancreatic duct and vessels. Total volume injected typically ranges from 0.2 ml to 0.6 ml. Follow with standard duct-to-mucosa pancreaticojejunostomy:
  * Tying down the posterior duct-to-mucosa sutures.
  * Placing and tying the anterior duct-to-mucosa sutures.
  * Tying down the posterior outer layer sutures.
  * Placing the anterior outer layer sutures. Meticulously avoid glue contact with sutures/mucosa Reconstruction: Complete the hepaticojejunostomy and duodenojejunostomy (or gastrojejunostomy).
  Other Names: NBCA
  Arms: N-butyl-2-cyanoacrylate (Histoacryl® )Injection Group.
Procedure: Standard Pancreaticojejunostomy — Patients randomized to this group will undergo pancreaticoduodenectomy and pancreaticojejunostomy using the standard surgical technique of the institution, without the application of N-Butyl-2-Cyanoacrylate or any other sealant to the pancreatic anastomosis. No placebo injection will be administered.
  Other Names: Standard PJ
  Arms: Standard Pancreaticojejunostomy

SUMMARY:
This randomized controlled trial investigates the safety and efficacy of injecting N-butyl-2- cyanoacrylate (Histoacryl®) into the pancreatic parenchyma during pancreaticoduodenectomy (PD) to enhance the security of the pancreaticojejunostomy (PJ) anastomosis and reduce postoperative pancreatic fistula (POPF) rates.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the efficacy of pancreatic parenchymal N-Butyl-2-Cyanoacrylate (NBCA) injection in reducing the incidence and severity of postoperative pancreatic fistula (POPF) after pancreaticoduodenectomy (PD). POPF remains a major complication of PD, leading to increased morbidity, mortality, and healthcare costs. NBCA, a tissue adhesive, has shown promise in various surgical applications due to its hemostatic and sealing properties. This study will enroll approximately 90 patients undergoing PD, randomly assigning them to either the NBCA injection group or the control group. The primary outcome will be the incidence of POPF according to the International Study Group on Pancreatic Surgery (ISGPS) definition. Secondary outcomes includes length of hospital stay, readmission rates, reoperation rates, mortality, and other postoperative complications. This trial is designed to provide high level evidence regarding the utility of NBCA in improving outcomes after PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreaticoduodenectomy for malignant lesions meeting the curative treatment intent in accordance with clinical guidelines.
* Soft pancreatic texture.
* Small main pancreatic duct diameter (<3 mm).
* Informed consent obtained.

Exclusion Criteria:

* Known hypersensitivity to cyanoacrylate or Lipiodol®.
* Extremely hard, fibrotic pancreas.
* Significant pancreatitis involving the pancreatic remnant.
* Active infection at the surgical site.
* Uncontrolled coagulopathy.
* Unfit patients for surgery due to severe medical illness.
* Inoperable patients with distant metastases, including peritoneal, liver, distant lymph node metastases, and involvement of other organs.
* Irresectable tumors in diagnostic laparoscopy.
* Patients requiring left, central or total pancreatectomy or other palliative surgery.
* Pregnant or breastfeeding women.
* Patients with serious mental disorders.
* Patients with vascular invasion and requiring vascular resection.
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative pancreatic fistula | Up to 90 days post-surgery
  A drainage fluid of any measurable volume with an amylase level more than three times the upper normal serum level on or after the 3rd postoperative day.

SECONDARY OUTCOMES:
Incidence of postoperative acute pancreatitis | 1 day post index surgery
  Altered serum amylase count on postoperative day 0 or 1
Incidence of Post-Pancreatectomy Hemorrhage | 90 days
  As defined by the International Study Group for Pancreatic Surgery (ISGPS), grade A, B and C rates
Incidence of intra-abdominal abscess | 90 days
  Collection containing gas bubbles, determining systemic signs of infection
Incidence of biliary fistula | 90 days
  Output of bile from drains on or by post operative day 3
Rate of readmission | 30 days after hospital discharge
  New admission within 30 days of discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Seewald S, Sriram PV, Naga M, Fennerty MB, Boyer J, Oberti F, Soehendra N. Cyanoacrylate glue in gastric variceal bleeding. Endoscopy. 2002 Nov;34(11):926-32. doi: 10.1055/s-2002-35312. No abstract available. PMID 12430080
- [Background] Lamsa T, Jin HT, Sand J, Nordback I. Tissue adhesives and the pancreas: biocompatibility and adhesive properties of 6 preparations. Pancreas. 2008 Apr;36(3):261-6. doi: 10.1097/MPA.0b013e31816714a2. PMID 18362839